CLINICAL TRIAL: NCT05395078
Title: Effects of Thoracic Extension Versus Thoracic Stabilization Exercises on Pain, Stiffness, Range of Motion, Disability and Posture in Patients With Maigne's Thoracic Pain.
Brief Title: Effects of Thoracic Extension Versus Thoracic Stabilization Exercises in Patients With Maigne's Thoracic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR &AHS/22/0134 Rubab
Record Dates: First submitted 2022-05-23; First posted 2022-05-27 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Thoracic
Keywords: Magnie's thoracic pain; Hyperkyphosis; Thoracic stabilization; Extension exercises
MeSH Terms: conditions — Kyphosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Thoracic extension exercises
  Interventions: Other: Conventional physical therapy treatment along with thoracic extension exercises
- Group B (Experimental): Thoracic Stabilization exercises
  Interventions: Other: Conventional physical therapy treatment along with thoracic stabilization exercises

INTERVENTIONS:
Other: Conventional physical therapy treatment along with thoracic extension exercises — Thoracic Extension Exercises (2 sets of 10 reps each/day). This exercise program will target thoracic spine extension and trunk muscle flexibility. A specialized program of thoracic extension in sitting, in prone lying, in quadruped position, on foam roller, wall angle stretch, corner stretch + hot pack (10 min) + Trapezius and Levator Scapulae stretching + Myofascial Release + Thoracic spinal mobilization (3 sets of 3 reps each/day). A total of 45 minutes session three times a week on alternate days for 3 weeks.
  Assessment will be done at baseline, on the end of 3rd week and for long term effects at the end of 6th week.
  Arms: Group A
Other: Conventional physical therapy treatment along with thoracic stabilization exercises — Thoracic Stabilization Exercises (2 sets of 10 reps each/day). This exercise program will target thoracic musculature, static and dynamic thoracic posture. A specialized program of Draw- in and chin tucks in crook lying, prone, sitting and standing, prone chin- tuck elevation exercises with arm at sides, arms behind head or overhead (4) + hot pack (10 min) + Trapezius and Levator Scapulae stretching + Myofascial Release + Thoracic spinal mobilization (3 sets of 3 reps each/day). A total of 45 minutes session three times a week on alternate days for 3 weeks. Assessment will be done at baseline, on the end of 3rd week and for long term effects at the end of 6th week.
  Arms: Group B

SUMMARY:
The aim of this study is to compare the effects of thoracic extension versus thoracic stabilization exercises on pain, stiffness, range of motion, disability and posture in patients with Maigne's thoracic pain.This study will be a randomized clinical trial and 32 patients fulfilling the inclusion criteria will be included in the study. they will be allocated into 2 groups using non- probability purposive sampling technique. Group A will receive conventional treatment, myofascial release, thoracic spine mobilization with Thoracic Extension exercise program, while Group B will receive conventional treatment, myofascial release, thoracic spine mobilization with Thoracic Stabilization exercise program. Outcome measure: Numeric Pain Rating Scale, Goniometer, Thoracic Stiffness Index, Revised Oswestry Thoracic Pain Disability Questionnaire, standing thoracic X-ray and Flexi curve ruler, will measure pain, thoracic flexion and extension, Cobb's angle, kyphosis index, thoracic stiffness index and disability. Both groups will receive a total of 45 minutes session, thrice a week for 3 weeks. Measurements will be taken at the baseline, at the end of 3rd week and for long-term effects at the end of 6th week. Data will be analyzed by SPSS version 21.

DETAILED DESCRIPTION:
Maigne's thoracic pain is a condition in which pain originates from the thoracic spine, but according to Maigne, in most cases, its origin lies in the lower three cervical segments. It is common among both men and women, but it is most common among women. Common symptoms of Maigne's thoracic pain are tenderness and stiffness of thoracic muscles, especially interscapular muscles. The most important and chief complaint reported by patients of this condition is unilateral and severe pain which increases with static sitting and with carrying or lifting heavyweight. Physical examination of tenderness on the interscapular region at the level of T5-T6, 1-2 cm lateral to the midline. Pressure reproduces the patient's pain. Several clinical trials have established therapeutic guidelines and protocols for the rehabilitation of hyperkyphosis. These trials have typically focused on the use of spinal bracing, therapeutic taping, manual therapy, and therapeutic exercise for postural training. Studies have been conducted on the effectiveness of combination therapy of thoracic extension exercises with other therapeutic exercises. Similarly, many studies have been conducted on thoracic stabilization exercises for posture correction. It is quite difficult to judge which exercise is more effective than the other. Moreover, typically for the management of Maigne's Thoracic pain, the efficacy of therapeutic treatment is quite underexplored. The rationale of this study is that it will provide evidence that may improve treatment strategies for the management of Maigne's Thoracic pain, majorly focusing on the muscular component of the thoracic region.

ELIGIBILITY:
Inclusion Criteria:

* Patients of age between 20-45 years
* NPRS value more than or equal to 4
* Cobb's Angle > 40°
* Chronic Maigne's Thoracic pain

Exclusion Criteria:

* Structural abnormalities
* Neoplasm
* Neurogenic problem
* H/o cervical or thoracic surgery
* H/o whiplash injury
* Muscular strain
* Lactating mothers
* Pregnant or 6 months post-partum females

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
NPRS | 3rd Week
  The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10) that best reflects the intensity of his/her pain 11-point numeric scale ranges from '0' representing no pain to 10 representing the worst imaginable pain
Goniometer | 3rd Week
  The science of measuring the joint ranges in each plane of the joint is called goniometry. Goniometer is a device that measures an angle or permits the rotation of an object to a definite position. Thoracic flexion and extension will be assessed through it.
Standing Thoracic X-ray | 3rd Week
  One lateral view X-ray of each subject will be taken of the thoracic spine at the hospital radiography department. Subjects will stand in a relaxed position with arms elevated in front of them for the X-ray. Cobb's angle will be measured from X-ray.
Kyphosis Index (KI) | 3rd Week
  Kyphosis Index will be measured using Flexi curve ruler, which is a flexible plastic 60-cm ruler to evaluate surface contour of thoracic curvature. The KI will be calculated by multiplying 100 by the value of thoracic width divided by thoracic length or KI = (thoracic width/length) ×100.
Thoracic Stiffness Index (TSI): | 3rd Week
  The TSI will be calculated as the value of the:
  KI in relaxed posture divided by the KI in best posture.
Revised Oswestry Thoracic Pain Disability Questionnaire (ROTPDQ) | 3rd Week
  It is a self-reported measurement tool that measures both pain and functional status and is used for evaluating disability caused by thoracic pain.

CONTACTS AND LOCATIONS:
Overall Officials: Syed Shakil-ur Rehman, Principal Investigator — Riphah International University
Locations (1):
- Riphah Rehabilitation Center, PSRD, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jain A, Srivastava D, Mishra A. Effects of targeted back muscle exercises in reducing thoracic kyphosis in patients of hyperkyphosis. International Journal of Orthopaedics. 2020;6(4):885-90.
- [Background] Almujel KN, Almhmd AE, Alharfy AAN, Albalawi IAS, Alanazi TBF, Alshehri AJ, et al. Causes and Management of Hyperkyphosis. Journal of Pharmaceutical Research International, July. 2021:1-8.
- [Background] Jang HJ, Hughes LC, Oh DW, Kim SY. Effects of Corrective Exercise for Thoracic Hyperkyphosis on Posture, Balance, and Well-Being in Older Women: A Double-Blind, Group-Matched Design. J Geriatr Phys Ther. 2019 Jul/Sep;42(3):E17-E27. doi: 10.1519/JPT.0000000000000146. PMID 28914720
- [Background] Dutton M, Magee D, Hengeveld E, Banks K, Atkinson K, Coutts F, et al. Orthopaedic examination, evaluation, and intervention: McGraw-Hill Medical; 2004.
- [Background] Pfeifer M, Begerow B, Minne HW. Effects of a new spinal orthosis on posture, trunk strength, and quality of life in women with postmenopausal osteoporosis: a randomized trial. Am J Phys Med Rehabil. 2004 Mar;83(3):177-86. doi: 10.1097/01.phm.0000113403.16617.93. PMID 15043351
- [Background] Bautmans I, Van Arken J, Van Mackelenberg M, Mets T. Rehabilitation using manual mobilization for thoracic kyphosis in elderly postmenopausal patients with osteoporosis. J Rehabil Med. 2010 Feb;42(2):129-35. doi: 10.2340/16501977-0486. PMID 20140408
- [Background] Greig AM, Bennell KL, Briggs AM, Hodges PW. Postural taping decreases thoracic kyphosis but does not influence trunk muscle electromyographic activity or balance in women with osteoporosis. Man Ther. 2008 Jun;13(3):249-57. doi: 10.1016/j.math.2007.01.011. Epub 2007 Apr 12. PMID 17433756
- [Background] Kang NY, Im SC, Kim K. Effects of a combination of scapular stabilization and thoracic extension exercises for office workers with forward head posture on the craniovertebral angle, respiration, pain, and disability: A randomized-controlled trial. Turk J Phys Med Rehabil. 2021 Sep 1;67(3):291-299. doi: 10.5606/tftrd.2021.6397. eCollection 2021 Sep. PMID 34870115
- [Background] Toprak Celenay S, Ozer Kaya D. An 8-week thoracic spine stabilization exercise program improves postural back pain, spine alignment, postural sway, and core endurance in university students:a randomized controlled study. Turk J Med Sci. 2017 Apr 18;47(2):504-513. doi: 10.3906/sag-1511-155. PMID 28425239
- [Background] Piri H, Hajian M, Mirkarimpour SH, Sheikhhoseini R, Rahimi M. The Effect of 12-Week Corrective Exercises on the Postural Angles of Beautician Females with Upper Crossed Syndrome: a Clinical Trial Study. Women's Health Bulletin. 2021:63-70.